CLINICAL TRIAL: NCT00314548
Title: Trial of Inhaled Alprostadil to Improve Hypoxia and Pulmonary Hypertension
Brief Title: Inhaled Prostacyclin for Adult Respiratory Distress Syndrome (ARDS) and Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Medical Research Council, Pakistan (Other)
Responsible Party: Dr. Shahla Siddiqui, Aga Khan University/Pakistan Medical Research Council
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-22-3/05/RDC/AKU/3479
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2009-11

CONDITIONS: Adult Respiratory Distress Syndrome; Pulmonary Hypertension
Keywords: ARDS; pulmonary hypertension; prostacyclins
MeSH Terms: conditions — Respiratory Distress Syndrome; Hypertension, Pulmonary | interventions — Alprostadil; Epoprostenol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cases (Experimental): PGE1 drug
  Interventions: Drug: PGE1 (prostacyclin)
- Placebo (Placebo Comparator): normal saline via same nebulizer
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: PGE1 (prostacyclin) — alprostadil nebulization
  Other Names: alprostadil
  Arms: Cases
Drug: normal saline — nebulize for 30 mins
  Arms: Placebo

SUMMARY:
Summary of the proposed research:

The intravenous application of prostacyclin (PGE1) or its stable analogue, iloprost, has been used to cause a decrease not only of the pulmonary but also of the systemic vascular tone. Aerosolized prostacyclin, on the other hand, can result in a selective pulmonary vasodilatation without affecting the systemic blood pressure as shown in preliminary studies/case reports. No large trials exist for this type of use of the drug so far. Furthermore, aerosolized PGI2 can improve gas exchange and pulmonary shunt in clinical settings of impaired ventilation/perfusion ratio as it occurs in adult respiratory distress syndrome (ARDS) due to the redistribution of pulmonary blood flow from non-ventilated to ventilated, aerosol accessible lung regions. Therefore, the investigators propose to carry out a prospective, double blinded, randomized trial to show that the nebulized iloprost decreases pulmonary hypertension selectively and improves oxygenation in ARDS.

DETAILED DESCRIPTION:
Introduction:

Pulmonary hypertension, defined as mean PA (pulmonary arterial) pressure of > 25 mm Hg, is an end point of a variety of conditions. These include primary pulmonary hypertension, post-operative pulmonary hypertension and as a result of increased pulmonary vascular resistance that occurs in ARDS. This is an entity distinguished by hypoxemia, non-cardiogenic pulmonary edema and bilateral infiltrates on chest X-ray. Prostacyclin (PGE1), an arachidonic acid metabolite, or its stable analogue, iloprost, has been evaluated for its efficacy in the treatment of pulmonary hypertension and for its use in reducing intra-pulmonary shunting in ARDS. While the intravenous application of iloprost can cause a decrease not only of the pulmonary but also of the systemic vascular tone, the aerosolized prostacyclin can result in a selective pulmonary vasodilatation without affecting the systemic blood pressure as demonstrated in preliminary studies/reports. Furthermore, aerosolized iloprost can improve gas exchange and pulmonary shunt in clinical settings of impaired ventilation/perfusion ratio as it occurs in ARDS, due to the redistribution of pulmonary blood flow from non-ventilated to ventilated, aerosol accessible lung regions.

Previous case reports and non-randomized studies have indicated that inhalation of aerosolized iloprost may offer a new life saving strategy in intractable pulmonary hypertension and ARDS. Further, advantages of inhaled iloprost include the lack of adverse reactions and toxic side effects as well as convenient and more cost-effective administration. Other available therapies like nitric oxide inhalation costs more, around Rs 350/liter and a total of 34-45 liters per patient is required. It is also associated with additional side effects, such as thrombocytopenia. Due to the irreversible nature of ARDS associated with high rate of mortality also affecting resource allocation in critically ill patients, we suggest carrying out this study in our intensive care unit (ICU), where the incidence is > 10% resulting in almost 90% mortality (ICU Quality Indicators Jan-Apr 20048). Iloprost is completely metabolized and excretion of metabolites is primarily via the kidneys; the elimination half-life is 30 minutes. Inhalation therapy reduces systemic absorption and hence elimination half-life.

In a previous study, aerosolized iloprost was found effective in improving the functional class of the patient, exercise capacity and improved shunting. However, large randomized trials are needed to prove the efficacy of this cost effective therapy in patients with pulmonary hypertension and ARDS.

Objectives:

To carry out a prospective, double blinded, randomized trial to show that the nebulized PGE1, a stable prostacyclin derivative, decreases pulmonary hypertension selectively and improves oxygenation in ARDS.

*ALPROSTADIL (20 mcg ampule) manufactured by Schering, Pakistan.

Importance of work:

Prostacyclin (PGE1), an arachidonic acid metabolite, has been evaluated for its efficacy in the treatment of pulmonary hypertension and for its use in reducing intra-pulmonary shunting in ARDS. While the intravenous application PGE1, or alprostadil, can cause a decrease not only of the pulmonary but also of the systemic vascular tone, the aerosolized PGE1 results in a selective pulmonary vasodilation without affecting the systemic blood pressure. Furthermore, aerosolized PGE1 can improve gas exchange and pulmonary shunt in clinical settings of impaired ventilation/perfusion ratio as it occurs in ARDS, due to the redistribution of pulmonary blood flow from non-ventilated to ventilated, aerosol accessible lung regions.

Critical review of relevant literature on the subject:

Previous case reports and non randomized studies have indicated that inhalation of aerosolized alprostadil may offer a new life saving strategy in intractable pulmonary hypertension and ARDS. Further, advantages of inhaled iloprost include the lack of adverse reactions and toxic side effects as well as convenient and more cost-effective administration. Due to the irreversible nature of ARDS associated with high rate of mortality also affecting resource allocation in critically ill patients, we suggest carrying out this study in our intensive care unit (ICU), where the incidence is > 10% resulting in almost 90% mortality (ICU Quality Indicators Jan-Apr 20048).

In a previous study, aerosolized alprostadil was effective in improving the functional class of the patient, exercise capacity and improved shunting. Large randomized trials are needed to prove the efficacy of this cost effective therapy in patients with pulmonary hypertension and ARDS. Other available therapies like nitric oxide inhalation costs higher around Rs 350/liter and a total of 34-45 liters per patient is required. It is also associated with additional side effects, such as thrombocytopenia.

Resume of any related work carried out by the principal investigator or co-Investigator in this area:

The principal investigator and co-investigator have the relevant qualification, experience and expertise to conduct this study, as is obvious from the list of recent selected publications.

Controls:

From selected patients included in the study in a random, blinded manner. Patients will be given a drug or placebo to be determined by pharmacy.

Work Up:

After enrolling, the following tests will be carried out to determine inclusion/ exclusion criteria.

* Transthoracic echo - to rule out ejection fraction < 30%
* Pulmonary embolus
* Pulmonary hypertension (TR jet) to be determined by echo
* Arterial blood gas
* CXR reviewed to determine ARDS criteria

Drug Administration:

Drug (alprostadil/placebo - normal saline) to be nebulized; 5 micrograms via standard nebulizer within 4 hours, once.

Standardization of Critical Care:

Standardization of treatment modalities have been incorporated in the methodology with regard to ventilatory support, inotropic support and fluid management; however, as the intensive care unit at the AKUH is an 'open unit' where patients are primarily taken care of by the primary teams and a critical care consultant (of which the PI is one), strict guidelines cannot be enforced. However we have given a general range of parameters, keeping in mind the recommendations of the Society of Critical Care medicine and the Acute Respiratory Distress Syndrome Network.

Once enrolled, the patients will be managed by the ICU consultant and the primary physician (may not always include PI). The following broad criteria will be followed in order to treat the patient:

1. Ventilatory support in ARDS/Pulmonary hypertension:

   * Any ventilatory mode can be used
   * Peak airway pressures (Pa) will be maintained under 35 mm Hg
   * Peep range to be between 8-14 mm Hg
   * Tidal volumes of 6 cc/kg
2. Inotropic Support:

   Dopamine (5-20 mics/kg/min) as a positive inotrope (dopaminergic, alpha and beta agonist activity) and norepinephrine (0.1-0.5 mics/kg/min) as a vasopressor (alpha agonist) are used for increasing blood pressure. The goal will be to maintain a mean arterial pressure (DBP plus 1/3 rd of pulse pressure) of > 60 mm Hg.
3. Fluid management:

Keeping a wedge pressure < 20 mm Hg will be the goal of fluid management.

Sample Size:

Assuming total Karachi population of over 150,000 (1998 Demographic Survey of Pakistan) of all age groups, and taking incidence of 20% (+/- 105 bound of error) of pulmonary hypertension and ARDS at 95% confidence interval, we extricated a sample size to be 91 cases (with 91 controls). Epi-info version 1.1 was used to calculate sample size. Actual sample size 182.

Outcome Measures:

* If met, trial will be terminated early in favor of using the drug. Positive result will be taken as PA pressures - mean PA pressure decreases by 10 in 4 hours and PaO2/FiO2 ratio - increases by 50 (or PaO2 increases by 10) in 4 hours.
* Results will be recorded in a Data Sheet - (see Appendix I).

Tests done: Arterial blood gases. Transthoracic echo before and after drug.

Ethics: Written approval of Aga Khan University Ethics Review Committee (ERC) has been obtained prior to commencement of the study.

Blinding: Each patient after enrollment will be assigned a serial number consecutively after meeting inclusion criteria reviewed by the principal investigator and research assistant. After the necessary workup and consent, drug shall be obtained from the AKUH pharmacy. The pharmacy will carry out randomization and deliver either alprostadil or normal saline (placebo) in an unmarked vial. Delivery dose and frequency will be carried out similarly for all patients. Data will be collected by the research assistant and nurse. At the end of the trial (after all cases and controls have been enrolled) the serial numbers of the patients will be matched to the delivery chart of the pharmacy to see whether they received the drug or placebo.

Year wise plan of work to be used during period:

All ICU patients.

Inclusion exclusion (Pulm. HTN, ARDS) (not intubated, no swan)

echo LVF, RVF, pulmonary embolus

Swan ganz catheter (wedge < 20)

consent (serial # and inform pharmacy)

ELIGIBILITY:
Inclusion Criteria:

After obtaining informed consent the following patients will be included:

* All patients admitted to the ICU with pulmonary hypertension (mean PA > 35 mmHg).
* All patients in ICU with post operative pulmonary HTN (mean PA > 35 mm Hg).
* All patients with ARDS (PaO2/FiO2 < 200 - arterial hypoxemia, bilateral infiltrates on Chest X-ray infiltrates on CXR and a wedge < 20 mm Hg on swan ganz parameters) or signs of heart failure.

Exclusion Criteria:

Patients to be excluded will be those with:

* Pulmonary embolus.
* Cor pulmonale.
* Ejection fraction of < 30%, wedge > 20 mm Hg.
* Non-intubated patients.
* Pediatric patients (< 16 yrs of age).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio increases by 10 | 30 mins

SECONDARY OUTCOMES:
PA [pulmonary artery] pressures decrease by 10 mm Hg | 30 mins

CONTACTS AND LOCATIONS:
Overall Officials: Shahla Siddiqui, MBBS, DABA, Principal Investigator — Aga Khan University

REFERENCES:
- [Background] 1. Domenighetti G, Stricker H. et al. Nebulized prostacyclin in ARDS: impact of primary and secondary disease on gas exchange response. Crit Care Med. 2001 ;29 (1) :57-62 2. Macherndl S, Kneussl M. et al. Long term treatment of pulmonary hypertension with aerosolized iloprost. Eur Respir J. 2001; 17(1): 8-13 3. Max M, Rossaint R. Inhaled prostacyclin in the treatment of pulmonary hypertension. Eur J Pediatr. 1999; 158 supp 1: S23-6. 4. Hoeper M, Olschewski H.et al. A comparison of the acute hemodynamic effects of inhaled nitric oxide and aerosolized iloprost in primary pulmonary hypertension. German PPH study group. J AM Coll Card. 2000 ; 35(1):176-82. 5. Olschewski h, Ghofrani H. et al. Inhaled iloprost to treat severe pulmonary hypertension. An uncontrolled trial. German PPH study group. Ann Int Med. 2000 21;132 (6):435-43.